CLINICAL TRIAL: NCT04009213
Title: A Multi-center, Randomized, Controlled, Single Blinded, Parallel-group Study Evaluating the Clinical Performance and Safety of LiquiBand FIX8® Versus Control for Hernia Mesh Fixation and Peritoneal Closure in Groin Hernia Repair
Brief Title: A Clinical Study to Evaluate the Clinical Performance and Safety of LiquiBand FIX8® Versus AbsorbaTack™ for Hernia Mesh Fixation and Peritoneal Closure in Groin Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LBF8-01 Version 1.3
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hernia; Inguinal Hernia; Femoral Hernia; Groin Hernia
Keywords: Laparoacopic; Peritoneal Closure
MeSH Terms: conditions — Hernia; Hernia, Inguinal; Hernia, Femoral

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two treatment arms, LiquiBand FIX8® or Control (AbsorbaTack™) device at a 1:1 ratio. Subjects will also be randomized according to laparoscopic technique used (TEP or TAPP hernia repair procedure), so that there is appropriate distribution between the Investigational and control devices. Randomization will occur immediately prior to use of either device for mesh fixation (TEP repairs) or mesh fixation and peritoneal closure (TAPP repairs only) and only after the Investigator has laparoscopically inspected the site of repair and determined the patient to be eligible for participation in the study.
Who Masked: Participant
Masking Description: Randomization to either Investigational or control device will occur at the surgery visit. The patients will be blinded to their randomly assigned treatment device prior to surgery and during the follow up period following surgery. While it is not possible to blind investigators/staff members to the treatment device used, Investigators and staff members will not learn of randomized device until immediately prior to use of device, so as to maintain subject blinding prior to the hernia repair. Investigators and staff members will be asked to maintain subject blinding through the course of the follow up visits so as to not bias subject feedback on applicable study assessments. Patients will receive the same standard of care prior to, during and following surgery regardless of randomized device assignment, and therefore will not be able to individually determine what device they have been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- LiquiBand FIX8® (Experimental): LiquiBand FIX8® is an n-butyl-2-cyanoacrylate adhesive monomer and D&C Violet #2 dye
  Interventions: Device: LiquiBand FIX8®
- AbsorbaTack™ (Active Comparator): AbsorbaTack™ is an absorbable synthetic polyester copolymer derived from lactic and glycolic acid and is dyed with D&C Violet No. 2
  Interventions: Device: AbsorbaTack™

INTERVENTIONS:
Device: LiquiBand FIX8® — An n-butyl-2-cyanoacrylate adhesive monomer and D&C Violet #2 dye
  Arms: LiquiBand FIX8®
Device: AbsorbaTack™ — An absorbable synthetic polyester copolymer derived from lactic and glycolic acid and is dyed with D&C Violet No. 2.
  Arms: AbsorbaTack™

SUMMARY:
This is a multi-center, randomized controlled trial of 284 subjects (142 in each group). Patients will be blinded to the fixation method used. The objective of this study is to compare the efficacy and safety of the LiquiBand FIX8® device to the tack-based control device (AbsorbaTack™) for laparoscopic groin hernia (inguinal or femoral) repair. The primary outcome measure is an improvement in pain score measured by VAS at 6 months. Secondary outcomes include the ability to affix hernia mesh, the ability to approximate the peritoneum, recurrence rate, and quality of life (Carolina Comfort Scale).

ELIGIBILITY:
Inclusion Criteria:

Is male or female, ≥22 years of age

Is willing and able to give written informed consent

Has a primary or recurrent groin hernia (unilateral or bilateral, inguinal or femoral)

Is currently scheduled and eligible for TAPP or TEP laparoscopic groin hernia repair (inguinal or femoral)

Hernia mesh to be used at the time of surgery is at least 4" x 6" in size and is one of the following;

* 3D Max™ Mesh (Bard Inc.)
* 3D Max™ Light (Bard Inc.)
* Parietex™ 2D (order code starting with TEC) Flat Sheet Mesh (Medtronic)
* Parietex™ 3D (order code starting with TET) Flat Sheet Mesh (Medtronic)

Is willing and able to comply with the protocol assessments at time of surgery and during the post surgical follow up period

Exclusion Criteria:

Has a hernia type not suitable for laparoscopic hernia repair as determined by the Investigator (i.e. strangulated)

Subject has a recurrent groin hernia previously repaired laparoscopically, has an anatomical defect or had prior surgical procedures that in the opinion of the Investigator prevents access to the pre-peritoneal space for TAPP or TEP laparoscopic hernia repair

Is pregnant or actively breastfeeding

Has a known sensitivity to cyanoacrylate or formaldehyde,D&C Violet No.2 dye or any component of LiquiBand FIX8® or control device

Has an active or potential infection at the surgical site or systemic sepsis

Hernia mesh to be used at surgery is less than 4"x6" in size, or not one of the types of mesh listed in Inclusion Criteria above

Cannot tolerate general anaesthesia

Has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Roth, Medicine, Principal Investigator — University of Kentucky College of Medicine
Locations (6):
- United States (6):
  - Cleveland Clinic, Weston, Florida
  - University of Kentucky College of Medicine UK Medical Center, Lexington, Kentucky
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Overlake Medical Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2019 and December 2021, 329 patients were screened and consented for laparoscopic groin (femoral and inguinal). Of those Subjects 142 were randomized to LiquiBand Fix8 and 142 were randomized to AbsorbaTack for mesh fixation and peritoneal closure (in the case of TAPP).
Groups:
- LiquiBand FIX8®: Subjects requiring laparoscopic (TEP and TAPP) hernia repair were randomized to LiquiBand FIX8®, for mesh fixation and peritoneal closure (in the case of TAPP).
- AbsorbaTack™: Subjects requiring laparoscopic (TEP and TAPP) hernia repair were randomized to AbsorbaTack™ for mesh fixation and peritoneal closure (in the case of TAPP).
Period: Overall Study
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Started | 142 | 142
Completed | 132 | 134
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Population: The analysis population n=284 Subjects, were randomized and enrolled into the investigational study and formed the ITT population.
Groups:
- LiquiBand FIX8®: Groin Hernia Study Arm with LiquiBand FIX8® as treatment
- AbsorbaTack™: Groin Hernia Study Arm with AbsorbaTack™ as treatment
- Total: Total of all reporting groups
Arm/Group | LiquiBand FIX8® | AbsorbaTack™ | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.41 (13.696) | 58.47 (14.411) | 58.94 (14.041)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 132 | 138 | 270
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 138 | 138 | 276
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall population differs for the AbsorbaTack™ group as n=1 patient did not provide a population description.
  Participants
    number analyzed (Participants) | 142 | 141 | 283
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 3 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 13 | 16 | 29
    White | 128 | 121 | 249
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 142 | 142 | 284

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Change in pain from baseline to 6 month will be assessed and compared to treatment with AbsorbaTack™ in subjects requiring laparoscopic (TEP and TAPP) hernia repair where the VAS value is 0 - 10, 0 = no pain and 10 = worst pain imaginable.
Time Frame: Assessed at pre-surgery (baseline), day 7, day 14, month 1, month 3 and month 6 post surgery. Change from baseline at month 6 reported.
Population: ITT population defined as all enrolled subjects. All patients for whom VAS measurements were recorded at Baseline and 6 month post surgery
Measure: Mean (Standard Deviation); unit: score on a VAS scale
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 136 | 133
score on a VAS scale | -4.9 (2.5) | -5.1 (2.3)
Statistical Analysis 1: Comparison: LiquiBand FIX8® vs AbsorbaTack™; Test type: Non-Inferiority — H0: δT - δC ≥ 0.9 Ha: δT - δC < 0.9; p < 0.025, ANCOVA

2. Secondary Outcome: Number of Participants With Hernia Recurrence
Description: The incidence of hernia recurrence was assessed by physical examination and confirmed by ultrasound imaging following physical examination. Also, the study sites were guided to ask the subjects 3 questions during the clinic visit performed remotely with a 'Yes' or 'No' response; 1. Do you think your hernia has come back? 2. Do you feel or see a bulge? and 3. Do you have physical pain or symptoms at the site?
Time Frame: Assessed at week 2, month 3, month 6 and month 12 post surgery. Month 12 post surgery reported
Population: ITT population defined as all enrolled subjects. All patients who attended their follow up visit and underwent a physical examination where possible, or alternatively with self-assessment for hernia recurrence.
Measure: Count of Participants; unit: Participants
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 141 | 140
Participants | 1 | 2
Statistical Analysis 1: Comparison: LiquiBand FIX8® vs AbsorbaTack™; Test type: Non-Inferiority — H0: qT - qC ≥ 10% H1: qT - qC < 10%; p < 0.025, Farrington-Manning

3. Secondary Outcome: Successful Mesh Fixation at the Time of Surgery.
Description: LiquiBand FIX8® was required to successfully fix hernia mesh at a rate non-inferior to control device (AbsorbaTack™). Successful mesh fixation did not require any additional fixation by alternate fixation device.
Time Frame: Time of surgery.
Population: All Subjects who underwent surgery with LiquiBand FIX8® or control
Measure: Count of Participants; unit: Participants
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 142 | 142
Participants | 142 | 142
Statistical Analysis 1: Comparison: LiquiBand FIX8® vs AbsorbaTack™; Test type: Non-Inferiority — H0: pC - pT ≥ 10% H1: pC - pT < 10%,; p < 0.025, Farrington-Manning

4. Secondary Outcome: Incidence of Successful Peritoneal Closure (TAPP Repairs Only)
Description: LiquiBand FIX8® was required to successfully approximate the peritoneum at a rate non-inferior to control device. Successful peritoneal closure did not require any additional fixation by alternate fixation device or additional procedure.
Time Frame: Time of surgery.
Population: ITT Population. Successful peritoneal closure at time of surgery was measured in all subjects undergoing TAPP hernia repair.
Measure: Count of Participants; unit: Participants
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 94 | 92
Participants | 82 | 84
Statistical Analysis 1: Comparison: LiquiBand FIX8® vs AbsorbaTack™; Test type: Non-Inferiority — H0: πC - πT ≥ 15% H1: πC - πT < 15%,; p < 0.025, Farrington-Manning

5. Secondary Outcome: Quality of Life as Measured by the Carolinas Comfort Scale (CCS).
Description: Quality of Life was assessed by completion of the Carolinas Comfort Scale (CCS) Questionnaire. CCS scores at each timepoint were compared between the LiquiBand FIX8® and control (AbsorbaTack) treatment groups. Carolinas Comfort Scale measures quality of life through a 23-item, Likert-type questionnaire that measures severity of pain, sensation of mesh and movement limitations in eight categories: laying down, bending over, sitting up, activities of daily living, coughing or deep breathing, walking, stairs and exercise. The subscales scores for pain (0-40), sensation of mesh (0-40) and movement limitations (0-35) are combined to provide a total CCS score. The best possible score is 0 and the worst possible score is 115.
Time Frame: Pre-Surgery, Week 1, Week 2, Month 1, Month 3, Month 6, Month 9 and Month 12 post surgery
Population: ITT population defined as all enrolled Subjects. All patients for whom a CCS questionnaire was completed prior to surgery and at 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months post surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 129 | 129
score on a scale
  Change from 1 week to 2 weeks | -7.7 (12.4) | -7.0 (13.2)
  Change from 1 week to 1 month | -12.4 (12.6) | -12.2 (14.6)
  Change from 1 week to 3 months | -14.6 (16.9) | -14.4 (15.9)
  Change from 1 week to 6 months | -15.1 (16.0) | -15.3 (16.7)
  Change from 1 week to 9 months | -15.6 (16.3) | -15.7 (16.5)
  Change from 1 week to 12 months | -15.6 (16.0) | -15.3 (16.1)

6. Secondary Outcome: Levels of Pain Experienced as Measured by Visual Analogue Scale (VAS).
Description: A Visual Analog Scale (VAS) was used as a measure of pain where the VAS value is 0 - 10, 0 = no pain and 10 = worst pain imaginable.
Time Frame: Evaluation of pain will be measured at pre-surgery, discharge (up to 3 days), Week 1, Week 2, Month 1, Month 3, Month 6, Month 9 and Month 12 post surgery
Population: ITT population defined as all enrolled subjects. All patients for whom VAS measurements were recorded at discharge, and at 1 week, 2 weeks, 1 month, 3 months, 6 months, 9 months and 12 months post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 142 | 142
score on a scale
  Change from pre-surgery to discharge | -0.3 (3.4) | -0.1 (3.5)
  Change from pre-surgery to 1 week | -1.5 (2.8) | -1.5 (3.1)
  Change from pre-surgery to 2 weeks | -2.8 (2.8) | -2.7 (2.9)
  Change from pre-surgery to 1 month | -3.2 (2.8) | -3.1 (3.1)
  Change from pre-surgery to 3 months | -3.6 (2.9) | -3.4 (3.1)
  Change from pre-surgery to 6 months | -3.6 (3.0) | -3.5 (3.1)
  Change from pre-surgery to 9 months | -3.7 (2.9) | -3.5 (3.0)
  Change from pre-surgery to 12 months | -3.6 (2.9) | -3.5 (3.1)

7. Secondary Outcome: Safety as Measured by the Incidence of Adverse Events.
Description: The number of all adverse events whether or not determined to be related to the LiquiBand FIX8® device or control device (AbsorbaTack™).
Time Frame: Intraoperatively, Discharge, Week 1, Week 2, Month 1, Month 3, Month 6, Month 9 and Month 12 post surgery
Measure: Number; unit: Adverse Events
Groups:
- AbsorbaTack™: Subjects requiring laparoscopic (TEP and TAPP) hernia repair were randomized to AbsorbaTack™, for mesh fixation and peritoneal closure (in the case of TAPP).
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
Number analyzed (Participants) | 142 | 142
Adverse Events | 114 | 157

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from time of randomization through 12 month follow up
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, user or other persons. A clinical occurrence means that it affects or might affect a patient's normal function.
Arm/Group | LiquiBand FIX8® | AbsorbaTack™
All-Cause Mortality (participants affected / at risk) | 1/142 | 0/142
Serious Adverse Events (participants affected / at risk) | 11/142 | 16/142
Other Adverse Events (participants affected / at risk) | 28/142 | 49/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LiquiBand FIX8® (N=142) | AbsorbaTack™ (N=142)
Atrial Fibrillation (Cardiac disorders) | 1 | 3
Haematoma (Injury, poisoning and procedural complications) | 0 | 2
Inguinal Hernia (Gastrointestinal disorders) | 1 | 2
Neuralgia (Nervous system disorders) | 2 | 0
Cerebro Vascular Accident (Vascular disorders) | 0 | 1
Cervical vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (General disorders) | 0 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Incisional Hernia (General disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Leiomyosarcoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Medical device site infection (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Prostate cancer metastatic (Reproductive system and breast disorders) | 1 | 0
Tooth Abcess (Infections and infestations) | 0 | 1
Urethral injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract injury (Injury, poisoning and procedural complications) | 0 | 1
Urosepsis (Renal and urinary disorders) | 0 | 1
Vomiting (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LiquiBand FIX8® (N=142) | AbsorbaTack™ (N=142)
Seroma (Injury, poisoning and procedural complications) | 19 | 25
Groin Pain (Injury, poisoning and procedural complications) | 4 | 14
Urinary Retention (Renal and urinary disorders) | 5 | 5
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04009213/Prot_SAP_001.pdf